CLINICAL TRIAL: NCT01488461
Title: Phenotypic and Genotypic Studies in Congenital and Early Onset Ataxias
Acronym: ATAXIC
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: NI 08034; AOM 09178 (Other: Assistance Publique)
Record Dates: First submitted 2011-12-06; First posted 2011-12-08 (Estimated); Last update posted 2015-06-15 (Estimated); Status verified 2015-06

CONDITIONS: Congenital Cerebellar Ataxias; Early-onset Cerebellar Ataxias
Keywords: Congenital cerebellar ataxias; Genetics; Gene ATCAY; Gene ABC7; Cerebellar atrophy
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Family Based
Biospecimen Retention: Samples With DNA — Blood sample
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- patients ataxic
  Interventions: Genetic: blood sample

INTERVENTIONS:
Genetic: blood sample — Blood sample will be analysed in order to check presence or not of mutation in ABC7, SLC9A6, GPR56, ATCAY.

SUMMARY:
Congenital ataxias (CA) are rare, non progressive diseases, characterized by psychomotor retardation, hypotonia followed by ataxia. The presence of the "molar tooth" on MRI allowed to define Joubert syndrome, a peculiar form of CA. Apart from this group, CA are mostly associated with cerebellar atrophy or hypoplasia without molar tooth on MRI. CA are a clinically as well as genetically heterogeneous group of diseases. Early-onset ataxias are progressive but may be difficult to distinguish from CA in the first years of the disease. To date, few genes responsible for CA have been identified: ABC7 (X-linked CA associated with sideroblastic anemia), SLC9A6 (X-linked CA associated with severe mental retardation, autism and epilepsy), GPR56 (CA associated with polymicrogyria), ATCAY (pure CA in Cayman isolate); the involvement of the ATCAY and ABC7 genes has never been assessed in a large cohort of CA patients.

Primary objective:

To assess the frequency of mutations of the ATCAY and ABC7 genes in patients affected with non Joubert congenital or early-onset ataxia.

Secondary objective:

To identify new loci and/or genes responsible for CA To further describe the clinical phenotype of the CA and to assess the frequency of the various clinical types (pure CA/CA associated with spasticity/ syndromic CA, congenital/early-onset CA, sporadic/familial CA).

To describe the clinical phenotype of CA related to mutations in one of analysed genes.

DETAILED DESCRIPTION:
All patients will be examined by a geneticist or a neuropediatric. All clinical data will be collected.

Strategy of the molecular study :

1. for all multiplex and consanguineous families a linkage analysis (loci ATCAY and ABC7 and others AC known genes) will be performed.
2. For all sporadic patients as well as linked multiplex and consanguineous families : sequencing of all coding exons of the gene ATCAY and others AC known genes.
3. For all sporadic male patients and linked families : sequencing of all coding exons of the gene ABC7.
4. For all patients with suggestive features : sequencing of all coding exons of the gene GPR56, VLDLR, NHE6 or other candidate gene.
5. In consanguineous families : linkage analysis using SNP-array and analysis of candidate genes present in the regions of extended homozygosity
6. linkage analysis in dominant families and analysis of candidate genes in the linked regions.
7. If a new AC locus is identified (using linkage or CGH array), this gene will be sequenced in all patients.

ELIGIBILITY:
Inclusion Criteria:

* Patient, child or adult, affected with a congenital or early-onset ataxia defined by:
* Neurological symptoms observed before age of 2 years.
* Non progressive cerebellar ataxia observed at the time of examination. Karyotype done or in progress

Exclusion Criteria:

* Metabolic disease
* Specific MRI malformations suggesting a peculiar entity : molar tooth (joubert syndrome), superior vermis dysplasia with cleft (Oligophrenin)
* Muscle weakness and elevated creatine phosphokinase (CPK)
* Clearly progressive ataxia.
* Absence of signature of the informed consent.
* Absence of affiliation to social security

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All types
Sampling Method: Non-Probability Sample
Enrollment: 165 (Actual)
Dates: Start 2012-01; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Percentage of the patients with a mutation in one of the analysed genes. | 1 day

SECONDARY OUTCOMES:
Percentage of patients with severe/moderate/mild/absent intellectual deficiency | 1 day
Percentage of patients with/without epilepsy/spasticity/extraneurological features and nature and frequency of MRI anomalies | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Lydie Burglen, PhD, Principal Investigator — Assistance Publique
Locations (1):
- Hôpital Trousseau, Service de Génétique, Paris, France